CLINICAL TRIAL: NCT02916836
Title: Effect of the Use of a Therapeutic Conciliation Document at the Outlet of Hospital, on the Emergency Use of Hospital Care in Patient Aged Over 75 Years Old.
Acronym: IATROMED
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawal of the associated centers
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-PREPS-01
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Iatrogenic Effect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With TDC sheet: Use of therapeutic drug conciliation sheet (TDC) by the hospital and transmitted to the family practitioner with other usual documentation
  Interventions: Other: therapeutic drug conciliation sheet (TDC)
- Without TDC Sheet: transmission of usual documentation only to the family practitioner
  Interventions: Other: No Use of therapeutic drug conciliation sheet (TDC)

INTERVENTIONS:
Other: therapeutic drug conciliation sheet (TDC) — Use of therapeutic drug conciliation sheet (TDC)
  Groups: With TDC sheet
Other: No Use of therapeutic drug conciliation sheet (TDC)
  Groups: Without TDC Sheet

SUMMARY:
The drug iatrogenesis represents an important public health problem. In the Iatromed project, we want to to assess a specific therapeutic drug conciliation sheet (TDC). This multicenter observational study is focus on 750 patients aged over 75 year old with polymedication. The main objective will be to determine if the use of the TDC, at the discharge of hospital, allows to reduce the number of use in emergency care within the two month after their hospital discharge

DETAILED DESCRIPTION:
The drug iatrogenesis represents an important public health problem with 5-10% of the grounds of hospitalization after age 65, and more than 20% after 80 years. Based on this observation, the health authority has proposed in 2011 the realization of therapeutic drug conciliation particularly in the elderly with multiple pathologies and multiple drugs. Taking into account the central role of the family practitioner in prescriptions, and the importance of coordination information such as output of hospitalization (vector of many malfunctions), we have achieved a therapeutic drug conciliation sheet (TDC) based primarily on the information needs by family practitioner after hospitalization of their patients. The issue of this study is to assess the interest for the use of a such TDC on the decrease in the rate of rehospitalization in the target population.

To do this, we are proposing a multicenter observational study. Randomization would be across the centres. The study would focus on 750 patients more of 75 with polymedication. The follow-up will last 6 months.

The main objective will be to determine if the use of the TDC, at the discharge of hospital, allows to reduce the number of use in emergency care within the two month after their hospital discharge. The first secondary objective will be identical to the main objective but rated at 6 months and the second secondary objective will be to assess the impact of the use of the TDC on overall mortality at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* age ≥75 years
* patients with a medical prescription, including at least three different allopathic molecules including at least a treatment in one of the following therapeutic classes:
* cardiovascular treatment: antiarrhythmics, antihypertensive drugs, anticoagulants and antiplatelet all classes
* treatment of the central nervous system: analgesics, benzodiazepines, antidepressants, hypnotic, antipsychotic drugs of all classes.

  * family practitioner identified
  * trusted personne identified
  * Hospital output project establishes

Exclusion Criteria:

* not speaking french patient
* short survival time

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patient aged over 75 years old
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
rate of patient who will have used hospital care in emergency | at least one time within the two month after their hospital discharge
  The use of hospital care in emergency is defined as a consultation in an emergency room and/or an emergency hospitalization.
  An emergency hospitalization is an hospitalization for which programing was made maximum 48h before the admission in hospital or clinic. The use will be documented by contact with the patient (or the support person if necessary) and his doctor. Here, it should be noted that deaths will be accounted for in the urgently use of to the hospital care regardless of the place of death. This in intended to take into account the possibility that a death may be related to a drug iatrogenic event for which the patient has not had time to resort to the hospital care in emergency.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, Principal Investigator — Centre Hospitalier Universitaire de Nice